CLINICAL TRIAL: NCT01879137
Title: Copeptin After Arginine Infusion for the Differential Diagnosis of the Polyuria-Polydipsia Syndrome ''The CARGO-Study''
Brief Title: Copeptin After Arginine Infusion in Polyuria-Polydipsia Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: CARGO 2013
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Healthy; Polyuria-polydipsia Syndrome
Keywords: Copeptin; Arginin stimulation test
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Serum EDTA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy adults
- Patients with a polyuria-polydipsia syndrome

SUMMARY:
the purpose of the study is to investigate whether arginine infusion is a new tool to differentiate patients with diabetes insipidus, primary polydipsia and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. No medication except hormonal contraception

Exclusion Criteria:

1. Evidence of any acute illness
2. Subjects refusing or unable to give written informed consent
3. Pregnancy
4. Any evidence of disordered drinking habits and diuresis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults Patients with polyuria-polydipsia syndrome
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Discriminative value of copeptin after arginine infusion in the differential diagnosis of polyuria-polydipsia syndrome. | up to 120 minutes after the Arginine infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland